CLINICAL TRIAL: NCT04876105
Title: Do Treatment Preferences Change According to the Duration of the Pain of the Patients With Low Back Pain?
Brief Title: Treatment Preferences in Patients With Low Back Pain
Status: Completed | Type: Observational
Sponsor: Pamukkale University (Other)
Responsible Party: Principal Investigator, Ayşe Ünal, PT., PhD., Pamukkale University
Other Study IDs: 24.11.2020/24
Record Dates: First submitted 2021-05-05; First posted 2021-05-06 (Actual); Last update posted 2022-01-27 (Actual); Status verified 2022-01

CONDITIONS: Low Back Pain
Keywords: low back pain; acute pain; subacute pain; chronic pain; treatment preference
MeSH Terms: conditions — Low Back Pain; Acute Pain; Chronic Pain

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Acute-subacute group: According to the duration of low back pain, it is classified as acute pain if it lasts less than a month, subacute pain if it lasts for 1-3 months.
  Interventions: Other: Assesment of treatment preference
- Chronic group: According to the duration of low back pain, it is classified as chronic pain if it lasts for more than 3 months.
  Interventions: Other: Assesment of treatment preference

INTERVENTIONS:
Other: Assesment of treatment preference — Multiple-choice survey questions were created by the researchers based on the studies in the literature regarding the pain and treatment preferences of the participants

SUMMARY:
Together with the guidance of health professionals try to obtain information from media, popular magazines and books and the internet regarding diseases and treatment methods in patients with low back pain with the development of technology. In parallel with this information which they obtained, they turn to different treatment methods. This study was carried on examining how pain duration affects treatment preferences in patients with low back pain.

ELIGIBILITY:
Inclusion Criteria:

* Individuals between the ages of 18-65 with complaints of low back pain and no communication problems were included in the study.

Exclusion Criteria:

* Individuals with any systemic, neurological and / or orthopedic disease diagnosed other than complaint of low back pain were excluded from the study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: A total of 155 individuals between the ages of 18-65 with complaints of low back pain, meeting the inclusion criteria and agreeing to participate in the study were included in the study.
Sampling Method: Non-Probability Sample
Enrollment: 155 (Actual)
Dates: Start 2020-11-25 (Actual); Primary Completion 2021-04-30 (Actual); Study Completion 2021-10-15 (Actual)

PRIMARY OUTCOMES:
Evaluation of treatment preferences | 5 minutes
  Multiple-choice survey questions were created by the researchers based on the studies in the literature regarding the pain and treatment preferences of the participants. In this survey, the patients were asked to state which of the treatment methods applied for low back pain they knew and which of these methods they preferred.

SECONDARY OUTCOMES:
Visual Analog Scale | 1 minute
  Pain intensity
Oswestry Disability Index | 5 minutes
  Disability caused by low back pain

CONTACTS AND LOCATIONS:
Locations (1):
- Pamukkale University, Denizli, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No